CLINICAL TRIAL: NCT01751425
Title: Phase I-II Study of Ruxolitinib (INCB18424) for Patients With Chronic Myeloid Leukemia (CML) With Minimal Residual Disease While on Therapy With Tyrosine Kinase Inhibitors
Brief Title: Ruxolitinib in Treating Participants With Chronic Myeloid Leukemia With Minimal Residual Disease While on Therapy With Tyrosine Kinase Inhibitors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Per PI Request. 2) No additional benefit was noted with the addition of Ruxolitinib.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0697; NCI-2018-01797 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0697 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Myelogenous Leukemia, BCR-ABL1 Positive in Remission; Minimal Residual Disease; Philadelphia Chromosome Positive, BCR-ABL1 Positive Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasm, Residual | interventions — Dasatinib; Imatinib Mesylate; nilotinib; ruxolitinib

STUDY DESIGN:
Intervention Model Description: This study was stopped early and did not go on to phase II.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TKIs, ruxolitinib) (Experimental): Participants receive commercially available TKIs (imatinib mesylate, nilotinib, or dasatinib) as they had been receiving during the last 6 months and ruxolitinib PO BID. Courses repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Drug: Imatinib Mesylate; Drug: Nilotinib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP57148B; Gleevec; Glivec; STI 571; STI-571; STI571
Drug: Nilotinib — Given PO
  Other Names: AMN 107 Base Form
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424

SUMMARY:
This phase I/II trial studies the side effects and best dose of ruxolitinib and to see how well it works in participants with chronic myeloid leukemia with minimal residual disease while on therapy with tyrosine kinase inhibitors. Ruxolitinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD) of the combination of ruxolitinib and a tyrosine kinase inhibitor (TKI) in patients with chronic myeloid leukemia (CML). (Phase I) II. To determine the clinical activity of the combination of ruxolitinib and a TKI in patients with CML in complete cytogenetic remission (CCyR) with minimal residual disease (MRD). (Phase II)

SECONDARY OBJECTIVES:

I. To determine the clinical activity of the combination of ruxolitinib and a TKI in patients with CML. (Phase I) II. To determine the safety of the combination of ruxolitinib and a TKI in patients with CML in CCyR with minimal residual disease. (Phase II) III. Determine the overall survival, event-free survival and survival free from transformation to accelerated and blast phase. (Phase I and II) IV. Determine the effect of therapy on bone marrow progenitors in clonogenic assays. (Phase I and II) V. Investigate the effect of therapy on molecular responses as assessed by genomic deoxyribonucleic acid (DNA) polymerase chain reaction (PCR). (Phase I and II) VI. Determine the effect of therapy on TKI-resistant quiescent leukemic Philadelphia chromosome (Ph)+ stem cells (CFSEmax/CD34+) by flow cytometric evaluation of activated Crkl and Jak2. (Phase I and II) VII. Assess the effect of therapy on self-renewal and/or survival of leukemic stem cells by fluorescence in situ hybridization (FISH) analysis on colonies. (Phase I and II) VIII. Assess ruxolitinib pharmacokinetics (PK) in preselected time intervals during co-administration of this agent with TKIs. (Phase I and II)

OUTLINE: This is a phase I, dose-escalation study of ruxolitinib followed by a phase II study.

Participants receive commercially available TKIs (imatinib mesylate, nilotinib, or dasatinib) as they had been receiving during the last 6 months and ruxolitinib orally (PO) twice daily (BID). Courses repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Philadelphia chromosome (Ph)-positive or BCR/ABL-positive CML (as determined by cytogenetics, FISH, or PCR).
* Patients must be on continuous TKI therapy for management of their CML. Any commercially available and FDA- approved TKI can be used, i.e., imatinib mesylate (IM), nilotinib (NIL) or dasatinib (DAS). Patients may be receiving TKI at entry in the frontline or salvage setting, including patients currently on imatinib after alpha-interferon failure or on dasatinib or nilotinib after failure to prior therapy including imatinib.
* Patients must have received the current TKI for at least 18 months and not have increased their dose in the last 6 months.
* For the phase I portion of the study, patients may be included without a CCyR provided they remain in chronic or accelerated phase CML and have at least a complete hematologic response (CHR). For the Phase II portion of the study patients must be in complete cytogenetic remission (CCyR), regardless of the stage of disease they had at the time they started therapy with TKI.
* Patients must have detectable BCR-ABL transcript levels meeting at least 1 of the following criteria: Patient has never achieved a major molecular response (MMR, as defined by a BCR-ABL/ABL =< 0.1% in the international scale (currently equivalent to 0.28 in the MD Anderson Cancer Center [MDACC] molecular diagnostic laboratory), and transcript levels have shown in at least 2 consecutive measures separated by at least 1 month to have increased by any value; or achieved a major molecular response which has been lost, with an interim increase in transcript levels by at least one-log, confirmed in two consecutive analyses separated by at least 1 month; or patient has received therapy for at least 2 years & lacks a sustained major molecular response; or patient has received therapy for at least 5 years and lacks a sustained complete molecular response (CMR, defined as transcript levels still detectable in the MDACC molecular diagnostic laboratory).
* Patients must not have had a known interruption of TKI therapy of greater than 21 consecutive days or for a total of 6 weeks in the 6 months prior to enrollment.
* Patients must be able to understand and sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the institutional policies.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
* Bilirubin < 2 x upper limit of normal (ULN) (unless associated with Gilbert's syndrome).
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 x ULN.
* Absolute neutrophil count (ANC) >= 1 x 10(9)/L.
* Platelets >= 100 x 10(9)/L.
* Serum creatinine < 1.5 mg/dL or creatinine clearance greater or equal than 60 cc/min as defined by the Cockcroft-Gault equation.
* Women of childbearing potential should be advised to avoid becoming pregnant while on therapy with ruxolitinib and for 30 days after the last dose and practice effective methods of contraception. Men should be advised not to father a child while receiving treatment with Ruxolitinib and for 30 days after the last dose. Effective methods of contraception for this study include barrier methods (e.g., condoms, diaphragm); spermicidal jelly or foam; oral, depo provera, or injectable hormonal contraceptives; intrauterine devices; tubal ligation; and abstinence.

Exclusion Criteria:

* For the phase I portion of the study, patients in blast phase. For the phase II portion of the study, patients in accelerated or blast phase.
* Patients receiving any other investigational agents.
* Patients who are pregnant or breast-feeding.
* Patients with clinically significant heart disease (New York Heart Association [NYHA] class III or IV).
* Patients with corrected QT (QTc) > 480 msec.
* Patients taking a potent CYP3A4 inhibitor that cannot be changed to an alternate drug.
* Known or suspected hypersensitivity to ruxolitinib.
* Patients with advanced malignant hepatic tumors.
* Patients with known active hepatitis B or C, or human immunodeficiency virus (HIV) infection.
* Patients with other medical conditions or concomitant medications that in the opinion of the principal investigator may interfere with the therapeutic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-07-24 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Residual disease as measured by polymerase chain reaction (PCR) (Phase II) | Up to 7 years
  It will be determined if the residual disease as measured by PCR can decrease by at least 1 log or become undetectable within 12 months from the start of study therapy. The proportion of patients with response after 12 months of treatment will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M. Kantarjian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT01751425/Prot_SAP_000.pdf